CLINICAL TRIAL: NCT06719323
Title: Long-term Effects of Family WISH Program for Adolescents With Congenital Heart Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chi-Wen Chen (Other)
Responsible Party: Sponsor-Investigator, Chi-Wen Chen, Professor, National Yang Ming Chiao Tung University
Organization: National Yang Ming Chiao Tung University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 202401204RINC
Record Dates: First submitted 2024-11-27; First posted 2024-12-05 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Heart Defects, Congenital
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: To ensure assessor blinding, different personnel conducted the interventions and outcome assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experimental group: a 12-week Family WISH program
- Comparison group (Sham Comparator): Comparison group: a family walking health education sheet received
  Interventions: Behavioral: Comparison group

INTERVENTIONS:
Behavioral: Family Walking Instruction with Support by Heart (Family WISH) program — Researchers will compare the 12-week Family WISH program, based on self-efficacy theory, to a comparison group receiving a family walking health education sheet to evaluate the long-term effectiveness of the Family WISH program.
Behavioral: Comparison group — a family walking health education sheet received
  Arms: Comparison group

SUMMARY:
The goal of this clinical trial is to learn the long-term effects of "Family Walking Instruction with Support by Heart" (Family WISH) on frailty state, quality of life and family functioning among adolescents with congenital heart disease (CHD).

Researchers will compare the 12-week Family WISH program, based on self-efficacy theory, to a comparison group receiving a family walking health education sheet to evaluate the long-term effectiveness of the Family WISH program.

Participants will:

* Walk with family members for 20-30 minutes daily, at least 5 times per week, totaling 150 minutes per week.
* Keep a diary to record the frequency of their walks and any symptoms experienced.
* Complete questionnaires at baseline, and at 6, 12, and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* being between 12 and 18 years old;
* having received a diagnosis of CHD by a physician before age 2;
* having received a diagnosis of CHD with New York Heart Association (NYHA) functional class I, II, or III;
* having parents or guardians who were able to communicate in Mandarin, and being able to communicate in Mandarin themselves;
* not having cognitive impairments, and;
* voluntarily signing informed consent forms.

Exclusion Criteria:

* undergoing heart transplant surgery within the past year;
* receiving cardiac catheterization intervention or open-heart surgery within the past 6 months;
* having CHD with NYHA functional class IV; and
* having other congenital diseases

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 104 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
frailty state | at baseline, and at 6, 12, and 24 weeks
  self-reported questionnaire completed

SECONDARY OUTCOMES:
quality of life and family functioning | at baseline, and at 6, 12, and 24 weeks
  self-reported questionnaires completed

CONTACTS AND LOCATIONS:
Locations (1):
- College of Nursing, National Yang Ming Chiao Tung University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No